CLINICAL TRIAL: NCT00911976
Title: Prospective Evaluation of the Xience V Everolimus-Eluting Stent In Saphenous Vein Graft Atherosclerosis: The Stenting Of Saphenous Vein Grafts Xience V Angiographic Study (SOS-Xience V)
Brief Title: Study of the Xience V Everolimus-eluting Stent in Saphenous Vein Graft Lesions
Acronym: SOS-Xience V
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: North Texas Veterans Healthcare System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Emmanouil Brilakis, Director, Cardiac Catheterization Laboratories, North Texas Veterans Healthcare System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 09-016
Record Dates: First submitted 2009-06-02; First posted 2009-06-03 (Estimated); Last update posted 2012-10-26 (Estimated); Status verified 2012-10

CONDITIONS: Coronary Artery Bypass; Atherosclerosis
Keywords: Coronary artery bypass; Stents; Angioplasty, Transluminal, Percutaneous Coronary; Coronary Restenosis; Everolimus; Saphenous vein grafts
MeSH Terms: conditions — Atherosclerosis; Coronary Restenosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Xience V (Experimental): Implantation of the Xience V stent in saphenous vein graft lesions
  Interventions: Device: Xience V coronary stent

INTERVENTIONS:
Device: Xience V coronary stent — The Xience V stent will be implanted in aortocoronary saphenous vein bypass graft lesions

SUMMARY:
The specific aim of the SOS-Xience V study is to examine the 12-month incidence of binary angiographic in-stent restenosis after implantation of the Xience V stent in aortocoronary saphenous vein bypass graft lesions.

DETAILED DESCRIPTION:
Implantation of bare metal coronary stents (BMS) is currently the preferred percutaneous treatment for aortocoronary saphenous vein bypass graft (SVG) lesions, but is associated with high risk for in-stent restenosis. Although drug-eluting stents (DES) appear promising, there are limited and conflicting data on their efficacy and safety in SVGs. Our group recently completed and reported the results of the SOS (Stenting Of Saphenous vein grafts) trial that compared a paclitaxel-eluting stent with a similar BMS. There is currently no data on the use of the second generation DES in these challenging lesions. The SOS-Xience V study will examine the effects of the Xience V everolimus-eluting stent in SVG lesions.

The specific aim of SOS-Xience V is to examine the 12-month incidence of binary angiographic in-stent restenosis (defined as a stenosis of > 50% of the minimum lumen diameter of the target segment) after implantation of the Xience V stent in SVG lesions.

The Xience V stent will be implanted in 40 consecutive patients who need stenting of a SVG lesion. Patients will undergo repeat follow-up angiography and intravascular ultrasonography at 12 months and will be followed clinically for 12 months to determine:

1. the incidence of binary angiographic in-stent restenosis, as assessed by 12 month follow-up quantitative coronary angiography (primary study endpoint), and
2. intra-stent intimal hyperplasia volume accumulation at 12 months, as measured by intravascular ultrasonography, and (b) 12-month incidence of ischemia-driven target vessel revascularization, stent thrombosis, and target vessel failure (composite of cardiac death, myocardial infarction, and target vessel revascularization) (secondary study endpoints), and (c) percent stent strut coverage by optical coherence tomography

ELIGIBILITY:
Inclusion Criteria:

1. Age > 18 years
2. Need for percutaneous coronary intervention of a 50-99% de novo SVG lesion that is between 2.5 and 4.5 mm in diameter, is ≤ 22 mm in length, and can be treated with implantation of a single stent
3. Use of an embolic protection device during the SVG intervention
4. Able and willing to return for angiographic follow-up after 12 months
5. Agree to participate and provide informed consent

Exclusion Criteria:

1. Use of stents other than the Xience V stent
2. Planned non-cardiac surgery within the following 12 months
3. Presentation with an ST-segment elevation acute myocardial infarction
4. Any previous percutaneous treatment of the target lesion (with balloon angioplasty, stent, intravascular brachytherapy etc)
5. Any previous percutaneous treatment of the target vessel (of a lesion different than the target lesion) within the prior 12 months
6. Hemorrhagic diatheses, or refusal to receive blood transfusions
7. Current treatment with warfarin
8. Recent positive pregnancy test, breast-feeding, or possibility of a future pregnancy
9. Coexisting conditions that limit life expectancy to less than 12 months
10. Patients who have a creatinine above 2.5 mg/dL (unless they require hemodialysis, in which case they are eligible to participate)
11. Patients allergic to contrast material that can not be adequately premedicated
12. History of an allergic reaction or significant sensitivity to everolimus
13. Documented left ventricular ejection fraction (LVEF) < 25% at most recent evaluation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2009-05; Primary Completion 2011-07 (Actual); Study Completion 2011-07 (Actual)

PRIMARY OUTCOMES:
the incidence of binary angiographic in-stent restenosis, as assessed by 12 month follow-up quantitative coronary angiography | 12 months

SECONDARY OUTCOMES:
intra-stent intimal hyperplasia volume accumulation at 12 months, as measured by intravascular ultrasonography | 12 months
incidence of ischemia-driven target vessel revascularization, stent thrombosis, and target vessel failure (composite of cardiac death, myocardial infarction, and target vessel revascularization) | 12 months
Percent stent strut coverage by optical coherence tomography | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Emmanouil S Brilakis, MD, PhD, Principal Investigator — North Texas Veterans Healthcare System; Subhash Banerjee, MD, Study Director — North Texas Veterans Healthcare System
Locations (1):
- VA North Texas Healthcare System, Dallas, Texas, United States

REFERENCES:
- [Result] Papayannis AC, Michael TT, Yangirova D, Abdel-Karim AR, Kohlhaas J, Mahmood A, Addo T, Haagen D, Makke L, Roesle M, Rangan B, Banerjee S, Brilakis ES. Optical coherence tomography analysis of the stenting of saphenous vein graft (SOS) Xience V Study: use of the everolimus-eluting stent in saphenous vein graft lesions. J Invasive Cardiol. 2012 Aug;24(8):390-4. PMID 22865309